CLINICAL TRIAL: NCT05881174
Title: Rapid Acupuncture Treatment for Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malcolm Grow Medical Clinics and Surgery Center (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Niemtzow, Lead Principal Investigator, Malcolm Grow Medical Clinics and Surgery Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20190055H
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: PTSD
Keywords: Acupuncture; PTSD; PCL-5 Questionnaire
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This is a 3 arm non-randomized, crossover-design clinical investigation using "rescue" acupuncture for the treatment of PTSD symptoms. Each patient receiving rescue acupuncture for PTSD will be their own "control."
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Newly untreated diagnosed PTSD patients without medications (Active Comparator): Newly untreated diagnosed PTSD patients who have not yet received any PTSD treatment for a 2-week therapy of acupuncture
  Interventions: Procedure: acupuncture
- Newly diagnosed PTSD patients on pharmacological therapy (Active Comparator): Newly diagnosed PTSD patients on pharmacological therapy for a 2-week therapy of acupuncture
  Interventions: Procedure: acupuncture
- Newly diagnosed PTSD patients with or without medications with mild traumatic brain injury (Active Comparator): Newly diagnosed PTSD patients with or without medications having mild traumatic brain injury for a 2-week therapy of acupuncture
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — acupuncture

SUMMARY:
The summary of this research study is to test the effectiveness of a rapid "rescue" acupuncture technique as a non-pharmacologic alternative treatment for the reduction of post-traumatic stress disorder (PTSD) symptoms in affected individuals as a means to improve warfighter health and enable a more rapid return to duty, especially in austere environments. Patients will receive acupuncture as a research-related course of treatment for PTSD. The PCL-5 questionnaire will be used to assess the presence and severity of PTSD symptoms. A PCL-5 questionnaire will be administered at the beginning of the first treatment of "rescue" acupuncture and after the last treatment. Following the acupuncture treatment, a PCL-5 questionnaire will be initiated at the beginning of the first week of treatment and the end of the second week of treatment at the participating Mental Health Clinic (pMHC).

DETAILED DESCRIPTION:
"The objective is to treat three ARMS of PTSD patients: ARM 1: Newly untreated diagnosed PTSD patients referred from a participating Mental Health Clinic (pMHC) who have not yet received any PTSD treatment for a 2-week therapy of ""rescue"" acupuncture (six 30 minute sessions Monday, Wednesday, and Friday); ARM 2: Newly diagnosed PTSD patients referred from the pMHC but already placed on pharmacological therapy (i.e. Prazosin, SSRI, sedative, etc.) prior to their enrollment in the pMHC; and ARM 3: newly diagnosed PTSD patients with or without medications referred to pMHC but have a mild traumatic brain injury that does not impede their judgment ability. ARMs 2 and 3 will follow the same ""rescue"" acupuncture program as ARM 1. A PCL-5 questionnaire will be administered prior to and after ""rescue"" acupuncture. ARMs 1, 2, and 3 patients will return to the pMHC (after 2 weeks of ""rescue"" acupuncture) to start or continue pharmacological and/or non-pharmacological therapy(s) and will also be evaluated by a PCL-5 questionnaire at the start and after 2 weeks. Statistical analysis of the PCL-5 questionnaire will compare the three ARMS together as to whether acupuncture is a benefit or not to the patient following therapies received for 2 weeks in the pMHC. The lowering of the PCL-5 symptomatic questionnaire score is a favorable indication of a benefit.

ELIGIBILITY:
Inclusion Criteria:

Active duty and retired military referred from a participating Mental Health Clinic

-

Exclusion Criteria:

Pregnancy Participated in a form of acupuncture in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
The Post Traumatic Stress Disorder Checklist (PCL-5) for the Diagnosis and Statistical Manual of Mental Disorders (DMS-5) Analysis | 6 Years
  Data will be analyzed using SAS v 9.4. The paired samples t-test will be used to assess the difference in PCL-5 score between pre and post acupuncture treatments. The paired samples t-test will be used to assess the difference in PCL-5 score between pre and post-pharmacological or non-pharmacological treatments. The ANOVA test will be used to assess differences in PCL-5 score between pharmacological, non-pharmacological or both pharmacological and non-pharmacological treatments. Mixed models will be used to assess differences in PCL-5 score between acupuncture treatments and pharmacological.
  The PCL-5 Analysis-pharmacological or both pharmacological and non-pharmacological treatment scale is a 20-item (0 = not at all, 4 = extremely) self-report measure that assesses the presence and severity of PTSD symptoms. The total severity score (min=0 and Max=80).
  A PCL-5 score of 31-33 or higher suggests the patient may benefit from PTSD treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Niemtzow, MD, PhD, MPH, Study Chair — Malcolm Grow Medical Clinics and Surgery Center; Songxuan Zhou Niemtzow, MD, LAc, Study Director — Malcolm Grow Medical Clinics and Surgery Center
Locations (1):
- Malcom Grow Medical Clinics and Surgery Center, Morningside, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data